CLINICAL TRIAL: NCT07193082
Title: Effect of Inspiratory Muscle Training on Diaphragm Muscle Thickness, Fatty Liver Density and Aerobic Capacity in Elderly Men: A Randomized Controlled Trial
Acronym: IMT AND ELDERL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gümüşhane Universıty (Other)
Responsible Party: Principal Investigator, Coşkun YILMAZ, ASSOC. PROF., Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025/0464
Record Dates: First submitted 2025-09-16; First posted 2025-09-25 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Aging; Inspiratory Muscle Weakness; Fatty Liver; Reduced Functional Capacity
Keywords: Aging; older women; exercise; gait; inspiratory muscle training; health
MeSH Terms: conditions — Fatty Liver; Motor Activity

STUDY DESIGN:
Intervention Model Description: Experimental (IMT Group): Inspiratory Muscle Training (POWERbreathe® device, twice daily, 30 breaths per session, 5 days/week, 4 weeks, resistance starting at 40% of MIP and increased weekly).
  Control Group: No inspiratory muscle training.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle training (Experimental): Experimental (IMT Group): Inspiratory Muscle Training (POWERbreathe® device, twice daily, 30 breaths per session, 5 days/week, 4 weeks, resistance starting at 40% of MIP and increased weekly).
  Interventions: Device: Experimental Inspiratory Muscle Training (IMT Group); Device: Control Group: No inspiratory muscle training.
- CONTROL (No Intervention): Control Group: No inspiratory muscle training.

INTERVENTIONS:
Device: Experimental Inspiratory Muscle Training (IMT Group) — Experimental (IMT Group): Inspiratory Muscle Training (POWERbreathe® device, twice daily, 30 breaths per session, 5 days/week, 4 weeks, resistance starting at 40% of MIP and increased weekly).
  Arms: Inspiratory muscle training
Device: Control Group: No inspiratory muscle training. — Control Group: No inspiratory muscle training.
  Arms: Inspiratory muscle training

SUMMARY:
This randomized controlled trial aims to investigate the effects of a 4-week inspiratory muscle training (IMT) program on diaphragm muscle thickness, fatty liver density, functional capacity, and quality of life in elderly men aged 60-80 years. Participants were randomized into an IMT group and a control group. Assessments included diaphragm thickness, fatty liver density (via CT), six-minute walk test (6MWT), and quality of life (SF-12).

DETAILED DESCRIPTION:
1. Introduction Modern lifestyles present a multitude of challenges, many of which differ markedly from those encountered by previous generations. The nature of these challenges has evolved over time, leading to significant shifts in the ways individuals maintain and protect their health. Consequently, primary health risk factors have also transformed. While the importance of preserving health to maintain quality of life is well established, the determinants influencing this process have undergone a substantial evolution. In contemporary contexts, the identification of key health determinants and the long-term monitoring of their effects have become essential for the development of effective health promotion strategies.

   Within this framework, physical activity and fitness have emerged as pivotal contributors to overall health and well-being in modern societies. Adequate levels of physical activity are positively correlated with favorable biomarkers and higher quality of life. This is particularly critical in aging populations, where maintaining physical activity levels supports functional capacity and mitigates age-related physiological decline.As aging progresses, health concerns such as sarcopenia, reduced muscle strength, and diminished functional capacity become increasingly prevalent.

   Respiratory muscle strength is especially affected by aging, declining by approximately 8-15% per decade after the age of 50, in both sedentary and active older adults. Muscle fiber counts in elderly individuals may decrease to only 20% of the total observed in young adults, and diaphragm and intercostal muscle strength can decline by up to 25% due to sarcopenia and muscle atrophy. This reduction in respiratory function can contribute to a decline in exercise tolerance and physical activity, thereby accelerating overall physiological deterioration. In this context, respiratory muscle function particularly diaphragm thickness serves as a key biomarker for ventilatory capacity and functional health in aging populations.

   Inspiratory muscle training (IMT) has gained increasing attention as a strategy to enhance functional capacity and support quality of life in both clinical and aging populations. However, prior research indicates that short-term protocols (e.g., 8 weeks) produce only modest and clinically insignificant improvements in maximal exercise capacity. In contrast, submaximal exercise assessments, such as the six-minute walk test (6MWT), better reflect daily functional activities and are therefore more suitable for evaluating clinically relevant improvements. This consideration informed the selection of 6MWT as a primary outcome in the present study.

   IMT exerts its physiological benefits primarily through delaying or attenuating the respiratory metaboreflex, thereby reducing respiratory fatigue, lowering blood lactate accumulation, and improving oxygen availability to locomotor muscles. It can induce adaptations such as diaphragm hypertrophy, enhanced respiratory efficiency, decreased dyspnea, improved endurance, favorable shifts in muscle fiber composition, and optimized neuromuscular control of respiratory muscles. Collectively, these mechanisms suggest that IMT has the potential to improve both functional performance and overall quality of life in aging adults, while potentially contributing to metabolic health by modulating factors such as fatty liver density. As the global population ages, international studies have emphasized the benefits of inspiratory muscle training (IMT) as a cost-effective and low-risk intervention for improving respiratory function, exercise performance, and quality of life in older adults.

   Based on this rationales, this study hypothesized that inspiratory muscle training would positively affect diaphragm muscle thickness, fatty liver, quality of life, and six-minute walk test performance in older men. In consideration of this hypothesis, the objective of this study was to examine the effect of inspiratory muscle training on diaphragm muscle thickness, liver fat percentage, quality of life, and 6-minute walk test (6MWT) performance in older men. A comprehensive evaluation of the relationships between these parameters, in conjunction with the comprehensive health benefits of IMT, may offer critical insights that facilitate the development of novel strategies to preserve functional independence and enhance quality of life in aging populations.
2. Materials and Methods 2.1. Participants This study was conducted as a parallel-group, pretest-posttest randomized controlled trial following the CONSORT guidelines. Before participation, all individuals received detailed information about the study and provided written informed consent following the ethical principles outlined in the Declaration of Helsinki. The study was designed following the principles of the Declaration of Helsinki and was approved by the Scientific Research Ethics Committee of Hitit University (meeting dated August 20, 2025, number 2025/5). This study aimed to investigate the effects of inspiratory muscle training (IMT) on diaphragm muscle thickness, abdominal wall thickness, and fatty liver density in man aged 60-80 years. The sample size was calculated using G*Power software (version 3.1.9.2) based on diaphragm thickness (DT) values reported in previous studies, with an alpha error of 0.05, a beta error of 0.2, and a medium effect size (f=0.25 or partial eta squared=0.06). Considering the study design, a dropout rate of approximately 50% was anticipated. Accordingly, a sample size of 20 participants (n = 10 per group) was initially determined. However, to minimize potential issues, it was decided to include a total of 30 participants by adding 50% more participants to each group.

2.2. Experimental design Men aged 60-80 years were invited to the laboratory on three separate occasions. During the first visit, participants were familiarized with the experimental procedures, and the IMT protocol was thoroughly explained and demonstrated. The second visit involved the collection of baseline (pre-training) measurements, including the six-minute walk test (6MWT), diaphragm thickness (DT), and fatty liver density (FLD), all assessed under the supervision of a radiologist. Following the completion of the four-week IMT training program, post-training measurements were obtained during the third visit 2.3. Liver Density Analysis In this study, data obtained from elderly man aged 60-80 years who underwent CT scanning of the thorax or abdomen for any clinical indication were used. Imaging was performed with a Siemens Somatom Definition AS 128 model computed tomography device. Participants were given breathing exercises before imaging. On the day of the imaging, the participants were placed on the device table in the supine position. After the device settings were completed, they were asked to take a deep breath and hold it just before the imaging started. Images were acquired in the inspiratory phase. In the acquired CT images, liver thickness was measured at a point with a relatively homogeneous thickness at the level of the liver dome in the posteromedial region of the right hemidiaphragm, and the data were recorded. Additionally, the density was measured in the same participants from a homogeneous parenchymal area without noticeable lesions in the segment eight region of the liver, adjacent to the middle hepatic vein, and the relevant data were recorded. As a result of the data, the device automatically calculated and recorded the liver fat content. A liver fat content value of less than 33 indicates more liver fat.

2.4. Diaphragm Thickness (DT) Measurement Diaphragm muscle thickness measurements were obtained from computed tomography images taken for clinical reasons. The GE Revo Evo Cardiac device (Revolution EVO, Revolution Maxima, Revolution Frontier, Revolution HD, Revolution CT, GE Healthcare, WI, USA) was used for imaging. A radiologist with expertise in thoracic computed tomography performed the measurements of diaphragm muscle thickness. During the imaging procedure, the subjects were in a supine position during the deep inspiration phase. Thickness measurements were obtained at the level of the upper pole of the right kidney. The measurements were taken perpendicular to the diaphragm axis, from the midline, and the posterior line of the vertebral body. At this juncture, the diaphragm muscle was visualised and its thickness was measured.

2.5. Body composition measurement The height of participants was measured to the nearest 0.1 centimetre using a standard height meter (Seca 769, Seca, Hamburg, Germany) while standing barefoot against a wall. Body weight was measured to the nearest 0,1 kilogram using a digital scale (Beurer, model GS27). Participants' body weight was measured in kilograms (kg) without shoes and while wearing shorts and a T-shirt to minimize the influence on the results.

2.6. Quality of Life Scale (QoL) Short Form-36 (SF-36) was developed by Ware et al. (1995) to measure quality of life. SF-12 Quality of Life Scale was formed by taking 12 different items from 8 subheadings of SF-36. Turkish validity and reliability study was conducted. In the scale, the functional status, well-being and general health perception of the individual are asked. Questions questioning physical and emotional status are answered as yes or no, and other questions include Likert-type options ranging between 3 and 6. Mental component summary (MCS) score is obtained from mental health, emotional role, social functioning and energy subcategories and physical component summary (PCS) score is obtained from physical role, physical functioning, general health and body pain subcategories. Scoring ranges from 0-100. A higher score is an indicator of better health. The calculation of sub-dimensions in the obtained data was made on https://orthopowertools.com/SF12.

2.7. Inspiratory muscle training (IMT) Inspiratory muscle training (IMT) was performed using the POWERbreathe® device (POWER® Breathe Classic, IMT Technologies Ltd., Birmingham, UK). The IMT protocol was administered twice daily, in the morning and evening, for four-week, with the intervention occurring five days per week. Each training session comprised 30 breathing cycles, with participants performing these exercises in the morning and evening, totaling 60 breathing cycles per day. Before using the POWERbreathe device, the resistance setting was calibrated to 40% of the participant's maximum inspiratory pressure (MIP), as reported in the study. The initial MIP value was increased by 10% every week. The training sessions were overseen by a certified trainer, who ensured that participants adhered to proper form. The morning IMT sessions were held between 8:00 a.m. and 10:00 a.m., and the evening sessions were held between 5:00 p.m. and 8:00 p.m.

2.8. Statistical analysis Statistical analyses were performed via SPSS (Version 21.0 for Windows, Chicago, IL, USA) software, with the statistical significance set at 0.05. The Shapiro-Wilk normality test was performed to determine the homogeneity of the sample. Repeated measures two-way analysis of variance and Bonferroni correction were used to analyze differences in fatty liver density, 6MWT, SF-12 and diaphragm thickness measurements between trials. Furthermore, the effect size in pairwise group comparisons was calculated using partial eta-squared (η p 2). The interpretation of the parameter η p 2 is as follows: small values, such as 0.01, indicate a small effect size; medium values, such as 0.06, indicate a medium-sized effect; and large values, such as 0.14, indicate a strong effect. The intraclass correlation coefficient (ICC) was calculated for the purpose of assessing the reproducibility of measurements obtained from the same observer. The interpretation of the results is as follows: scores between 0.50 and 0.75 are considered moderate, scores between 0.75 and 0.90 are considered good, and scores of 0.90 and above are considered excellent.

ELIGIBILITY:
Inclusion:

* Male, aged 60-80 years
* Healthy, without severe comorbidities
* Voluntary participation with informed consent

Exclusion:

* Known respiratory or cardiovascular disease
* Neurological or musculoskeletal disorders limiting participation
* Recent abdominal or thoracic surgery
* Inability to comply with training protocol

Ages: 60 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-06-05 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
fatty liver density | 4 weeks.
  Change in fatty liver density (CT measurement) from baseline to 4 weeks.
Diaphragm thickness | 4 weeks.
  Change in diaphragm thickness (CT measurement) from baseline to 4 weeks.

SECONDARY OUTCOMES:
6MWT distance | 4 weeks.
  Change in functional capacity (6MWT distance) after 4 weeks.
SF-12 Physical and Mental Component Scores | 4 weeks
  Change in health-related quality of life (SF-12 Physical and Mental Component Scores) after 4 weeks.
  The SF-12 health-related quality of life scale consists of 12 questions and assesses an individual's overall health-related quality of life in two main dimensions:
  Physical Component Summary (PCS) Covers subdomains such as physical functioning, limitations in daily activities, role limitations due to physical health, pain, and general health perception.
  Higher scores indicate better physical health and functioning. Mental Component Summary (MCS) Covers subdomains such as mental health, role limitations due to emotional problems, social functioning, and vitality/energy.
  Higher scores indicate better mental health and social well-being.
  Scoring:
  Scores are typically transformed into a 0-100 scale; some studies use norm-based scoring (mean 50 ± 10).
  Scores above 50 indicate above-average quality of life, while scores below 50 suggest lower quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Gumushane Univetsity, Gümüşhane, Kelkit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF